CLINICAL TRIAL: NCT05482971
Title: A Single-arm, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Ropeginterferon Alfa-2b-njft (P1101) in Adult Patients With Essential Thrombocythemia
Brief Title: A Single-arm, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of P1101 in Adults With ET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXCEED ET / A22-301
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Essential Thrombocythemia
Keywords: MPN; Myeloproliferative; Neoplasms; Myeloproliferative Neoplasms; Essential; Thrombocythemia; Besremi; Ropeginterferon Alfa-2b-njft; P1101; Essential Thrombocythemia
MeSH Terms: conditions — Thrombocythemia, Essential; Neoplasms; Myeloproliferative Disorders; Thrombocytosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ropeginterferon alfa-2b (P1101) (Experimental): Pre-filled Syringe, Q2W, SC injection
  Interventions: Drug: Ropeginterferon alfa-2b-njft (P1101)

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b-njft (P1101) — Ropeginterferon alfa-2b-njft (P1101)
  Other Names: P1101

SUMMARY:
A Single-arm, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Ropeginterferon alfa-2b-njft (P1101) in Adult Patients with Essential Thrombocythemia

DETAILED DESCRIPTION:
PharmaEssentia is developing a pegylated (PEG) IFN-α product, P1101, for the treatment of Essential Thrombocythemia (ET) as lack of disease modifying therapies in essential ET constitutes a serious issue in modern hematology.

Ropeginterferon alfa-2b-njft (P1101) may represent an effective, well-tolerated treatment with the ability to provide a deeper response and superior control of important blood parameters with the potential to alter the course of the disease and prevent progression to post-ET myelofibrosis (MF) and/or secondary acute myeloid leukemia (sAML). Ropeginterferon alfa-2b-njft (P1101) is currently being evaluated in comparison to ANA in the ongoing global Phase 3 clinical study, SURPASS ET.

Enrolled patients will receive P1101 over 13 months followed by an extension period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years old.
2. Subjects diagnosed with ET according to the World Health Organization (WHO) 2016 criteria.
3. Subjects that are cytoreductive treatment-naïve, or pre-exposed to HU and/or ANA, as specified below (according to Investigator's judgment and documented in the patient's medical record):

   a. Cytoreductive-naïve patients must be in need of cytoreductive treatment, defined as having at least one of the following:

   i. Progressive leukocytosis and/or thrombocytosis

   ii. Disease-related symptoms (i.e., pruritus, night sweats, fatigue)

   iii. Vasomotor/microvascular disturbances, not responsive to aspirin (including headache, chest pain or erythromelalgia, etc.)

   iv. High-risk (history of thrombosis at any age; or age >60 years with JAK2 mutation)

   b. Patients previously exposed to HU will be classified as either:

   i. Documented formal HU resistance or intolerance

   ii. HU stopped without documented formal resistance/intolerance due to insufficient blood count control or toxicity. The last HU dose must be >7 days prior the first dose of P1101.
4. Adequate hepatic function defined as bilirubin ≤1.5 × upper limit normal (ULN), prothrombin time (PT) (international normalized ratio, [INR]) ≤1.5 x ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 x ULN, aspartate aminotransferase ≤2.0 x ULN at screening.
5. Creatinine clearance ≥40 mL/min (by Cockcroft-Gault equation).
6. Males and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 60 days following the last dose of the study drug, and females must agree to not breastfeed during the study.
7. Written informed consent obtained from the subject and ability for the subject to comply with the requirements of the study.
8. Platelet count >450 × 109/L at screening
9. Both ANA-naïve and ANA-pretreated subjects are eligible for the study, regardless of the reason to terminate ANA use

Exclusion Criteria:

1. Any subject requiring a legally authorized representative
2. Subjects who stopped prior interferon alfa therapy due to low efficacy or poor tolerability
3. Any contraindications or hypersensitivity to IFN-α and/or its excipients
4. Co-morbidity with severe or serious condition that, in the Investigator's opinion, would jeopardize the safety of the subject or their compliance with the protocol, including significant cardiac disease (including New York Heart Association Class III-IV congestive heart failure and clinically significant arrhythmias) and pulmonary hypertension
5. History of major organ transplantation
6. Pregnant or lactating females
7. Subjects with any significant medical conditions that, in the opinion of the Investigator, would compromise the results of the study or may impair compliance with the requirements of the protocol, including but not limited to:

   1. Documented autoimmune disease at screening or in the history (e.g., thyroid dysfunction, hepatitis, idiopathic thrombocytopenic purpura, scleroderma, psoriasis, or any arthritis of autoimmune origin)
   2. Clinically relevant pulmonary infiltrates, pneumonia, and pneumonitis at screening that, in the Investigator's opinion, would jeopardize the safety of the subject or their compliance with the protocol
   3. Infections with systemic manifestations (e.g., bacterial, fungal, or human immunodeficiency virus [HIV], except hepatitis B [HBV] and/or hepatitis C [HCV],at screening)
   4. Evidence of severe retinopathy (e.g., cytomegalovirus retinitis [CMV], macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension)
   5. History or presence of clinically relevant depression
   6. Previous suicide attempts or at any risk of suicide at screening, in the judgment of the Investigator
   7. History or presence of clinically significant neurologic diseases
   8. History of any malignancy within 5 years (except adequately treated nonmelanoma skin cancer, prostate cancer status post resection with an undetectable prostate-specific antigen [PSA], curative treated in-situ cancer of the cervix, ductal carcinoma in-situ [DCIS] of the breast, Stage 1 Grade 1 endometrial carcinoma, or other solid tumors including lymphomas [without bone marrow involvement] curatively treated with no evidence of disease for ≥2 years prior to study)
   9. History of alcohol or drug abuse within the last year
   10. History or evidence of any other MPN
8. Use of any investigational drug <4 weeks prior to the first dose of study drug or not recovered from effects of prior administration of any investigational agent
9. Presence of more than one driver mutation (e.g., V617F JAK2 and CALR, CALR and MPL, V617F JAK2 and MPL)
10. Prior use of JAK inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess efficacy of ropeginterferon alfa-2b-njft (P1101) in adult USA/Canadian patients with ET | 12 months
  Efficacy will be based on peripheral blood count remission as defined by hematocrit (HCT) <45%, white blood cell (WBC) count ≤10 × 109/L, and platelets (PLT) ≤ 400 × 109/L in at least 80% of bi-weekly measurements for a consecutive 32-wek period during the 52-week core study treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Oleh Zagrijtschuk, MD, PhD, Study Director — PharmaEssentia Corporation
Locations (34):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Marin Cancer Care, Greenbrae, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The Winship Cancer Institute Emory University, Atlanta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine - Division of Oncology, St Louis, Missouri
  - Cancer Care Specialists, Reno, Nevada
  - Astera HealthCare, East Brunswick, New Jersey
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina (UNC) - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia - Emily Couric Cancer Center, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (4):
  - University of Calgary Tom Baker Cancer Centre, Calgary, Alberta
  - St. Paul's Hospital - Providence Health Care, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masarova L, Reeves BN, El Chaer F, Foltz L, Tashi T, Abu-Zeinah G, Lucas J, Halpern AB, Maze D, Qin A, Safah H, Lan F, O'Connell CL, Goel S, Rein L, Fang B, How J, Babu S, Li Z, Cerquozzi S, Oh ST, Hunter AM, Podoltsev N, Vachhani P, Yacoub A, Cunningham JM, Hillis C, Otoukesh S, Zagrijtschuk O, Castro H, Bose P. A multicenter study to assess efficacy, safety, and tolerability of ropeginterferon alfa-2b-njft in patients with essential thrombocythemia in the US and Canada: EXCEED-ET trial. Front Med (Lausanne). 2025 Apr 17;12:1548590. doi: 10.3389/fmed.2025.1548590. eCollection 2025. PMID 40330782